CLINICAL TRIAL: NCT01574937
Title: A Dose Finding Clinical Trial of Cabozantinib (XL 184) Administered in Combination With Abiraterone in Castration Resistant Prostate Cancer
Brief Title: XL-184+Abiraterone in Post-Chemo CRPC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Christopher Sweeney, MBBS, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-441
Record Dates: First submitted 2012-04-08; First posted 2012-04-10 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Prostate Cancer
Keywords: Castration Resistant; Post Chemotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cabozantinib; abiraterone; Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment Arm (Experimental): Cabozantinib and abiraterone
  Interventions: Drug: Cabozantinib; Drug: Abiraterone

INTERVENTIONS:
Drug: Cabozantinib — 28 day cycle
  Other Names: XL 184
Drug: Abiraterone — 28 day cycle
  Other Names: Zytiga

SUMMARY:
This research study is a Phase I clinical trial. Phase I clinical trials test the safety of an investigational drug. Phase I studies also try to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drug is still being studied and that research doctors are trying to find out more about it. It also means that the FDA (U.S. Food and Drug Administration) may not have approved this drug for use in participants, including people with your type of cancer.

In this research study, we are testing the safety of XL184 at different dose levels. XL184 is a new study drug, which is taken by mouth. Laboratory studies have shown that XL184 may prevent tumor growth by stopping the formation of blood vessels inside the tumor and also shrink tumors.

This drug has been used in early-stage studies and is also currently being studied in other trials. Information from those other research studies suggests that XL184 may help to slow or stop tumor growth including prostate cancer. We will also be taking blood and urine tests to look at how your body processes the drug.

DETAILED DESCRIPTION:
The following procedures will be performed during this study. On Day 1 for every cycle (28 days/4 weeks)-The following will be undertaken prior to initiating study therapy and on day 1 of every subsequent cycle: A medical history, physical exam, performance status, blood tests, urine test.

Since we are looking for the highest dose of the study drug that can be administered safely without severe or unmanageable side effects in participants, not everyone who participates in this research study will receive the same dose of the study drug. The dose you get will depend on the number of participants who have been enrolled in the study before you and how well they have tolerated their doses.

We will actively monitor your condition for up to 30 days after you come off the study. If you come off study for a side effect we will monitor your condition until the resolution or stabilization of the side effect

ELIGIBILITY:
Inclusion Criteria:

* CRPC with up to 2 prior chemotherapy regimens
* Progressive disease on CT, MRI or bone scan per mRECIST
* Has recovered to baseline/CTCAE less than or equal to Grade 1 from toxicities related to prior treatment (except alopecia)
* Agree to use accepted barrier method of contraception

Exclusion Criteria:

* Cytotoxic chemotherapy within 3 weeks
* Prior treatment with cabozantinib or other c-MET inhibitor
* Prior therapy with a lyase inhibitor
* Concurrent use of hormonal therapies other than LHRH analogue or orchiectomy
* Received radiation therapy to thoracic cavity or GI tract within 3 months, to bone or brain metastasis within 2 weeks or to any other site within 4 weeks of first dose of study drug
* Prior treatment with a small molecular kinase inhibitor within 2 weeks of study entry
* Received another investigational product within 28 days prior to study entry
* Active brain metastases or epidural disease
* Requires concomitant treatment in therapeutic doses with warfarin or warfarin-related agents
* No uncontrolled significant intercurrent or recent illness

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-04-03 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | 2 years
  To define the MTD of cabozantinib in combination with abiraterone

SECONDARY OUTCOMES:
Definition of a Dosing Regimen | 2 years
  To define a dosing regimen of abiraterone and cabozantinib suitable for further evaluation based on long term toxicity and efficacy data

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sweeney, MBBS, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No